CLINICAL TRIAL: NCT01699841
Title: Breast Milk Composition and HIV-exposed/Unexposed Early Infant Growth and Infectious Disease Events
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 1111002616
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: HIV; Malnutrition; Cryptosporidiosis
MeSH Terms: conditions — Malnutrition; Cryptosporidiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV+ and HIV- mothers and their infants

SUMMARY:
The purpose of this study is to understand how breast milk may protect infants from infection and promote favorable immunological, growth and development outcomes. By following mothers and their infants, we will evaluate the important interactions between infant immune responses and infectious disease events in relation to breast milk composition and feeding patterns. Our aim is to identify a set of predictive factors corresponding to healthy early infant growth and development in this setting in Northern Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by mothers, and parental consent on behalf of their infants
* Confirmed maternal HIV status (HIV-1, HIV-2 or HIV-Dual seropositive or HIV-seronegative)
* Stated intention to remain in the clinic catchment area ≥6 months post-partum
* Singleton birth

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV+ and HIV- mothers and their infants attending a semi-rural clinic and/or rural dispensaries from birth to 6 months of infant age in north western Tanzania.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2013-06-15 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Breast milk composition | Up to 6 months post-partum

SECONDARY OUTCOMES:
Infant anthropometric measures | Up to 6 months of age
Infant infectious disease events | Up to 6 months of age

CONTACTS AND LOCATIONS:
Locations (1):
- Kisesa Health Centre, Kisesa, Tanzania